CLINICAL TRIAL: NCT01452165
Title: Observational Study on Cardiac Morphology and Function in Patients With Peripheral Artery Disease in Vastmanland County, Sweden(PADVa).
Brief Title: Peripheral Artery Disease in Vastmanland
Acronym: PADVa
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Collaborators: Västmanland County Council, Sweden (Other Government)
Responsible Party: Sponsor
Other Study IDs: PADVa
Record Dates: First submitted 2011-10-11; First posted 2011-10-14 (Estimated); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Peripheral Vascular Diseases; Heart Failure; Ventricular Dysfunction
Keywords: Cardiovascular diseases; Hypertrophy, Left ventricle; Echocardiography; Prognosis
MeSH Terms: conditions — Peripheral Vascular Diseases; Heart Failure; Ventricular Dysfunction; Cardiovascular Diseases; Hypertrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and serum.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The main purposes of this study are:

* to describe the prevalence and degree of reduced left ventricular function and hypertrophy in patients with peripheral arterial disease in comparison to controls from the general population,
* to evaluate factors of importance to left ventricular dysfunction and hypertrophy in patients with peripheral arterial disease, and
* to assess the impact of cardiac function and left ventricular hypertrophy on long-term prognosis in patients with peripheral artery disease.

DETAILED DESCRIPTION:
Left ventricular dysfunction is often a consequence of coronary heart disease (CHD). CHD is prevalent among patients with peripheral artery disease. However, there is limited data regarding left ventricular morphology and function in those patients. In the cross-sectional part of this study we will describe the prevalence of reduced cardiac function and left ventricular hypertrophy in a cohort of patients with peripheral artery disease. The patient outcomes will be compared to control subjects randomly selected from the general population in a case-control design. Further, clinical and genetic determinants of cardiac dysfunction in the patient cohort will be identified. In the longitudinal part of the study, the impact of cardiac function and morphology on cardiovascular mortality and morbidity will be evaluated in the cohort.

ELIGIBILITY:
Inclusion Criteria:

Fulfillment of at least one of the following criteria:

* ankle-brachial-index (ABI) <= 0.9, or
* stenosis of > 30% of the internal carotid artery, or
* symptoms typical for claudication and corresponding stenotic findings on the ultrasound examination.

Exclusion Criteria:

* age less than 18 years
* severly impaired communication capabilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients referred to the Ultrasound laboratory of the Vascular Surgery Department for evaluation of known or suspected vascular disease.
Sampling Method: Probability Sample
Enrollment: 457 (Actual)
Dates: Start 2006-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Left ventricular ejection fraction (cross-sectional outcome measure) | baseline
  LVEF obtained by echocardiographic biplane disk summation method. In the cross-sectional study, the mean value of LVEF and the prevalence of reduced LVEF (LVEF < 50%) in the patient group will be compared to the control group.
Cardiovascular events (longitudinal outcome measure) | 5-10 years
  Cardiovascular events obtained from the Swedish National Causes of Death register and the Swedish National In-patient register. The registers are linked to the patients by the unique personal identification number assigned to each swedish resident.
Left ventricular mass (cross-sectional outcome measure) | baseline
  Left ventricular mass obtained by 2-dimensional echocardiography according to the American Society of Echocardiography.

SECONDARY OUTCOMES:
Wall motion score index (WMSI) | baseline
  Left ventricular wall motion score according to the American Society of Echocardiopgraphy.
Echocardiographic left ventricular filling variables | baseline
  Echocardiographic variables for evaluation of left ventricular diastolic function (e.g. E/A- and E/e'-ratios).

CONTACTS AND LOCATIONS:
Overall Officials: Pär Hedberg, Assoc. Professor, Study Chair — Center of Clinical Research, Uppsala university, Central Hospital, SE-72189 Västerås, Sweden; Jerzy Leppert, Senior Professor, Principal Investigator — Center of Clincial Research, Uppsala university, Central Hospital, SE-72189 Västerås, Sweden
Locations (1):
- Center of Clinical Research, Uppsala university, Central Hospital, Västerås, Sweden

REFERENCES:
- [Result] Hedberg P, Hammar C, Selmeryd J, Viklund J, Leppert J, Hellberg A, Henriksen E. Left ventricular systolic dysfunction in outpatients with peripheral atherosclerotic vascular disease: prevalence and association with location of arterial disease. Eur J Heart Fail. 2014 Jun;16(6):625-32. doi: 10.1002/ejhf.95. Epub 2014 Apr 26. PMID 24771615
- [Result] Hysing P, Jonason T, Leppert J, Hedberg P. Prevalence and prognostic impact of electrocardiographic abnormalities in outpatients with extracardiac artery disease. Clin Physiol Funct Imaging. 2018 Sep;38(5):823-829. doi: 10.1111/cpf.12488. Epub 2017 Nov 24. PMID 29171136
- [Result] Nowak C, Carlsson AC, Ostgren CJ, Nystrom FH, Alam M, Feldreich T, Sundstrom J, Carrero JJ, Leppert J, Hedberg P, Henriksen E, Cordeiro AC, Giedraitis V, Lind L, Ingelsson E, Fall T, Arnlov J. Multiplex proteomics for prediction of major cardiovascular events in type 2 diabetes. Diabetologia. 2018 Aug;61(8):1748-1757. doi: 10.1007/s00125-018-4641-z. Epub 2018 May 24. PMID 29796748
- [Derived] Dahle N, Arnlov J, Leppert J, Hedberg P. Nondipping blood pressure pattern predicts cardiovascular events and mortality in patients with atherosclerotic peripheral vascular disease. Vasc Med. 2023 Aug;28(4):274-281. doi: 10.1177/1358863X231161655. Epub 2023 Apr 10. PMID 37036102